CLINICAL TRIAL: NCT00713674
Title: Comparison of Decolonization of MRSA Using Theraworx
Brief Title: Comparison of Decolonization of Methicillin-resistant Staphylococcus Aureus (MRSA) Using Theraworx
Acronym: SJMRSA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patient recruitment.
Sponsor: Mercy Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SJMRSA-01
Record Dates: First submitted 2008-07-07; First posted 2008-07-11 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Methicillin-Resistant Staphylococcus Aureus
Keywords: Methicillin resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): No Treatment
- 2 (Experimental): Theraworx intranasal
  Interventions: Other: Theraworx
- 3 (Active Comparator): mupirocin antibiotic ointment intranasal
  Interventions: Drug: mupirocin antibiotic ointment

INTERVENTIONS:
Other: Theraworx — Theraworx swab intranasal BID for 5 days
  Arms: 2
Drug: mupirocin antibiotic ointment — mupirocin antibiotic ointment swab intranasal BID for 5 days
  Arms: 3

SUMMARY:
The purpose of this study is to examine treatment method of Methicillin-resistant Staphylococcus aureus (MRSA) decolonization in patients.

DETAILED DESCRIPTION:
Decolonization therapy is indicated for management of patients with MRSA. Theraworx is reported to be an effective antimicrobial against multiple organisms. In this study, patients with positive MRSA colonization culture will be treated with Theraworx to evaluate decolonization duration capability.

ELIGIBILITY:
Inclusion Criteria:

* Positive MRSA culture

Exclusion Criteria:

* Patients currently on or start antibiotic therapy directed for MRSA.(Prophylaxis antibiotic for surgical procedure not considered therapy.)
* Patients with MRSA infected wounds
* Patients under the age of 18 years
* A woman currently pregnant or nursing a child
* Patients participating in another study within 30 days of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Evidence of decolonization confirmed by intranasal culture | Up to 14 days post treatment (+/- 1-2 days)

SECONDARY OUTCOMES:
Economic-Cost comparison of treatment Evidence of decolonization | 5 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roger E Huckfeldt, MD, Principal Investigator — Mercy/St. John's Hospital - Springfield